CLINICAL TRIAL: NCT05938309
Title: A Prospective, Multicenter Cohort Study on the Efficacy and Safety of Laparoscopic Resection of 5cm or Larger Gastric Gastrointestinal Stromal Tumors
Brief Title: A Cohort Study on the Safety of Laparoscopic Resection of 5cm or Larger Gastric Gastrointestinal Stromal Tumors
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University (Other)
Collaborators: Fujian Provincial Hospital (Other); Fujian Cancer Hospital (Other Government); First Affiliated Hospital of Fujian Medical University (Other); 900 Hospital of Joint Logistics Support Force of PLA (Other); The First Affiliated Hospital of Xiamen University (Other); The Second Affiliated Hospital of Fujian Medical University (Other); The First Hospital of Putian City (Unknown); The Affiliated Hospital(Group) of Putian University (Unknown); Zhangzhou Municipal Hospital of Fujian Province (Other); Longyan City First Hospital (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Head of Department of Gastric Surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Other Study IDs: FUGES-029
Record Dates: First submitted 2023-06-19; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrectomy; Laparoscopic; gastrointestinal stromal tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- large group: laparoscopic resection of 5cm or larger gastric gastrointestinal stromal tumors
- small group: laparoscopic resection of less than 5cm gastric gastrointestinal stromal tumors

SUMMARY:
The purpose of this study is to explore the safety of laparoscopic resection of 5cm or larger gastric gastrointestinal stromal tumors

DETAILED DESCRIPTION:
There is a lack of high-quality evidence on the efficacy and safety of laparoscopic resection of gastric GIST over 5cm. A multicenter, prospective cohort study was conducted to evaluate the clinical efficacy of laparoscopic resection of 5cm or larger gastric gastrointestinal stromal tumors (GIST) compared to laparoscopic resection of GIST of less than 5cm. The primary evaluation parameter is overall postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years < age < 75 years
2. Primary gastric lesion diagnosed as gastric GSIT by endoscopic biopsy histopathology or suspected gastric GIST by preoperative endoscopy, ultrasound endoscopy, or CT or MR, and confirmed as primary gastric GIST by postoperative pathology
3. Patient informed consent and willingness to undergo laparoscopic resection
4. Expected laparoscopic outcome of R0 resection
5. Performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2, Preoperative American Society of Anesthesiologists（ASA） score I-III

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of upper abdominal surgery (except the history of laparoscopic cholecystectomy)
4. History of gastric surgery (except ESD/EMR for gastric cancer)
5. History of other malignant diseases within the past five years
6. History of unstable angina or myocardial infarction within the past six months
7. History of a cerebrovascular accident within the past six months
8. History of continuous systematic administration of corticosteroids within one month
9. Requirement of simultaneous surgery for other diseases
10. Emergency surgery due to complications (bleeding, obstruction, or perforation) caused by gastric cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are assigned to undergo gastrectomy for gastric gastrointestinal stromal tumors are included.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall postoperative morbidity | 30 days after surgery or the first discharge ( if over 30 days hospital stay)
  This is for the incidence of early postoperative complications, which defined as the event observed within 30 days after surgery.

SECONDARY OUTCOMES:
intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
Conversion to open surgery rate | 1 day
  Conversion to open surgery rate is defined as the rate of open surgery whatever the reason
Positive surgical margin rate | 1 day
  Positive surgical margin rate
The variation of white blood cell count | Preoperative 7 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of hemoglobin | Preoperative 7 days and postoperative 1, 3, and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 7 days and postoperative 1, 3, and 5 days
  The values of C-reactive protein in milligram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response
overall postoperative serious morbidity rates | 30 days after surgery or the first discharge ( if over 30 days hospital stay)
  According to the Clavien-Dindo complication scoring system, grade IIIA and above is a serious complication, and when multiple complications occur at the same time, the complication with the highest grade will prevail.
Time to first ambulation | 30 days
  Time to first ambulation in days is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year disease free survival rate | 36 months
  3-year disease free survival rate
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into four categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, and mixed type

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastric Surgery， Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joensuu H, Hohenberger P, Corless CL. Gastrointestinal stromal tumour. Lancet. 2013 Sep 14;382(9896):973-83. doi: 10.1016/S0140-6736(13)60106-3. Epub 2013 Apr 24. PMID 23623056
- [Background] Dematteo RP, Gold JS, Saran L, Gonen M, Liau KH, Maki RG, Singer S, Besmer P, Brennan MF, Antonescu CR. Tumor mitotic rate, size, and location independently predict recurrence after resection of primary gastrointestinal stromal tumor (GIST). Cancer. 2008 Feb 1;112(3):608-15. doi: 10.1002/cncr.23199. PMID 18076015
- [Background] Bischof DA, Kim Y, Dodson R, Carolina Jimenez M, Behman R, Cocieru A, Blazer DG 3rd, Fisher SB, Squires MH 3rd, Kooby DA, Maithel SK, Groeschl RT, Clark Gamblin T, Bauer TW, Karanicolas PJ, Law C, Quereshy FA, Pawlik TM. Open versus minimally invasive resection of gastric GIST: a multi-institutional analysis of short- and long-term outcomes. Ann Surg Oncol. 2014 Sep;21(9):2941-8. doi: 10.1245/s10434-014-3733-3. Epub 2014 Apr 24. PMID 24763984
- [Background] De Vogelaere K, Hoorens A, Haentjens P, Delvaux G. Laparoscopic versus open resection of gastrointestinal stromal tumors of the stomach. Surg Endosc. 2013 May;27(5):1546-54. doi: 10.1007/s00464-012-2622-8. Epub 2012 Dec 12. PMID 23233005
- [Background] Goh BK, Goh YC, Eng AK, Chan WH, Chow PK, Chung YF, Ong HS, Wong WK. Outcome after laparoscopic versus open wedge resection for suspected gastric gastrointestinal stromal tumors: A matched-pair case-control study. Eur J Surg Oncol. 2015 Jul;41(7):905-10. doi: 10.1016/j.ejso.2015.04.001. Epub 2015 Apr 15. PMID 25913060
- [Background] von Mehren M, Randall RL, Benjamin RS, Boles S, Bui MM, Casper ES, Conrad EU 3rd, DeLaney TF, Ganjoo KN, George S, Gonzalez RJ, Heslin MJ, Kane JM 3rd, Mayerson J, McGarry SV, Meyer C, O'Donnell RJ, Pappo AS, Paz IB, Pfeifer JD, Riedel RF, Schuetze S, Schupak KD, Schwartz HS, Van Tine BA, Wayne JD, Bergman MA, Sundar H. Gastrointestinal stromal tumors, version 2.2014. J Natl Compr Canc Netw. 2014 Jun;12(6):853-62. doi: 10.6004/jnccn.2014.0080. PMID 24925196
- [Background] Goh BK, Chow PK, Chok AY, Chan WH, Chung YF, Ong HS, Wong WK. Impact of the introduction of laparoscopic wedge resection as a surgical option for suspected small/medium-sized gastrointestinal stromal tumors of the stomach on perioperative and oncologic outcomes. World J Surg. 2010 Aug;34(8):1847-52. doi: 10.1007/s00268-010-0590-5. PMID 20407770
- [Background] Piessen G, Lefevre JH, Cabau M, Duhamel A, Behal H, Perniceni T, Mabrut JY, Regimbeau JM, Bonvalot S, Tiberio GA, Mathonnet M, Regenet N, Guillaud A, Glehen O, Mariani P, Denost Q, Maggiori L, Benhaim L, Manceau G, Mutter D, Bail JP, Meunier B, Porcheron J, Mariette C, Brigand C; AFC and the FREGAT working group. Laparoscopic Versus Open Surgery for Gastric Gastrointestinal Stromal Tumors: What Is the Impact on Postoperative Outcome and Oncologic Results? Ann Surg. 2015 Nov;262(5):831-9; discussion 829-40. doi: 10.1097/SLA.0000000000001488. PMID 26583673
- [Background] Khoo CY, Goh BKP, Eng AKH, Chan WH, Teo MCC, Chung AYF, Ong HS, Wong WK. Laparoscopic wedge resection for suspected large (>/=5 cm) gastric gastrointestinal stromal tumors. Surg Endosc. 2017 May;31(5):2271-2279. doi: 10.1007/s00464-016-5229-7. Epub 2016 Sep 8. PMID 27631317
- [Background] Park SH, Lee HJ, Kim MC, Yook JH, Sohn TS, Hyung WJ, Ryu SW, Kurokawa Y, Kim YW, Han SU, Kim HH, Park DJ, Kim W, Lee SI, Cho H, Cho GS, Kim JJ, Kim KH, Yoo MW, Yang HK. Early experience of laparoscopic resection and comparison with open surgery for gastric gastrointestinal stromal tumor: a multicenter retrospective study. Sci Rep. 2022 Feb 10;12(1):2290. doi: 10.1038/s41598-022-05044-x. PMID 35145127